CLINICAL TRIAL: NCT02212847
Title: Spatial Orientation and Vestibular Function in Patients With Acute or Chronic Unilateral Vestibular Deficits and in Patients With Bilateral Vestibular Deficits
Brief Title: Spatial Orientation and Vestibular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: vest_loss_percept_zurich
Record Dates: First submitted 2014-07-02; First posted 2014-08-08 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Vestibular Perception; Damaged Vestibular System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vestibular stimulation (Experimental)
  Interventions: Other: vestibular stimulation

INTERVENTIONS:
Other: vestibular stimulation

SUMMARY:
Spatial orientation is achieved through central integration of various sensory inputs and prior knowledge in a statistically optimal way based on the reliability of the different signals. When upright, the subjective visual vertical (SVV) is accurate and precise in healthy human subjects. However, when roll-tilted, both systematic physiologic, roll-angle dependent errors (termed A- und E-effect) and a decrease in precision of SVV estimates have been described. In case of a sudden unilateral vestibular deficit (UVD) a significant imbalance between the two vestibular organs occurs at the level of the vestibular nuclei, disrupting the percept of vertical. The most frequent cause for such a unilateral vestibular deficit is an inflammation of the vestibular nerve by viral infection, termed vestibular neuritis (VN). While in the acute stage these patients are usually immobilized due to the severity of symptoms, recovery is overall good and most patients return to their daily activities within a few weeks. Central compensation is considered the most important contributor to recovery in these patients, while recovery of the damaged vestibular nerve occurs only in a minority of cases. While acute VN presents with sudden UVD, bilateral vestibular deficits (BVD) typically evolve more slowly and re-sult in distinct complaints.

The percept of vertical can be quantified by assessing the subjective visual vertical or SVV, which is usually done by letting subjects adjust a luminous line along perceived direction of gravity. Modifications of this paradigm which are independent from retinal input are e.g. adjustments of a rod along perceived vertical in complete darkness (termed subjective haptic vertical or SHV) and self-alignments along perceived vertical (subjective postural vertical or SPV) and perceived horizontal (subjective postural horizontal or SPH) in complete darkness. Previous research has proposed no unified percept of vertical as errors assessed in different domains (visual, haptic, postural) were diverging in patients with acute UVD. While errors were profound for the SVV, the SPV remained accurate.

Here the investigators aim to quantify verticality perception in patients with either acute or chronic UVD and patients with BVD both in upright and roll-tilted positions. Specifically, the investigators will use different paradigms to address the ques-tion whether there is a unified percept of vertical and how a bias in this percept changes over time.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-75
2. informed consent
3. for group 1: acute (i.e. symptom onset less than 72 hours ago) unilateral vestibular deficit as confirmed by clinical examination (pathologic head-impulse test, no skew deviation, no gaze-evoked nystagmus).
4. for group 2: chronic (i.e. symptom onset more than 4 weeks ago) unilateral vestibular deficit as confirmed by vestibular testing in the acute stage (either abnormal unilateral response on caloric irrigation or video-head-impulse testing).
5. for group 3: chronic (i.e. symptom onset more than 4 weeks ago) bilateral vestibular deficits as confirmed by vestibular testing (bilaterally reduced response on caloric irrigation or video-head impulse testing).
6. absence of exclusion criteria

Exclusion Criteria:

1. History of a peripheral-vestibular deficit (valid only for group 4 - controls)
2. Disturbed consciousness
3. Personal history of traumatic brain injury, cerebrovascular disorders, seizures
4. History of chronic neck complaints including severe neck pain.
5. Alcohol dependency
6. Intake of anxiolytic, antidepressant, neuroleptic or sedative medication
7. Other neurological or systemic disorder which can cause cerebellar deficits, dementia, cognitive dysfunction, visuospatial or tactile neglect, aphasia or visual field deficits
8. Pregnancy or possible pregnancy if not ruled out by a negative pregnancy test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-07; Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
accuracy of verticality perception - baseline and change over 3 months | at baseline for the control group (while on the turntable over 1 hour) and change from baseline to follow-up after 3 months for the acute vestibular loss group (again over 1 hour)
  The accuracy of verticality perception is defined as the individual median value of a series of line adjustments along perceived direction of gravity (units: degrees). this results in a report of the participants perceived direction of gravity relative to true earth-vertical. Repetitive adjustments will be collected while on the turntable, each adjustment lasting up to 15seconds.

SECONDARY OUTCOMES:
precision of verticality perception - baseline and change over 3 months | at baseline for the control group (while on the turntable for 1 hour) and change from baseline to follow-up after 3 months for the acute vestibular loss group (again over 1 hour while on the turntable)
  The precision of verticality perception is defined as the individual median absolute deviation of single line adjustments along perceived direction of vertical (units: degrees). Repetitive adjustments will be collected while on the turntable, each adjustment lasting up to 15seconds. The resulting value reflects the amount of trial-to-trial variability in a given subject, which is inverse correlated to the precision.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Straumann, Prof MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No